CLINICAL TRIAL: NCT05452148
Title: Emergence of Specific Genotypes/Phenotypes of Pneumocystis Jirovecii in Solid Organ Transplant Recipients: Potential Involvement of Mycophenolic Acid
Brief Title: Specific Genotypes/Phenotypes of Pneumocystis Jirovecii in Solid Organ Transplant Recipients: Potential Involvement of Mycophenolic Acid
Acronym: IMPDH
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: IMPDH ( 29BRC22.0106)
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Transplantation; Pulmonary Diseases
Keywords: Pneumocystis jirovecii; IMPDH; Genetic variant
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Pneumocystis DNA isolates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the presence of IMDPH mutants of Pneumocystis jirovecii in solid organ transplant recipient with prior exposition to mycophenolic acid.

DETAILED DESCRIPTION:
Mycophenolic acid (MPA) targets inosine 5'-monophosphate dehydrogenase (IMPDH) of human lymphocytes. It is used as an immunosuppressant to prevent rejection in solid organ transplant (SOT) recipients who are otherwise at risk for Pneumocystis pneumonia (PCP). We recently hypothesized that MPA exerts selective pressure on Pneumocystis given the in vitro antifungal activity of this drug on other fungi. In a single center study, we identified a missense mutation G1020A in the impdh gene, corresponding to an amino acid change Ala261Thr in IMPDH protein, among Pneumocystis isolates from MPA-treated SOT recipients. Considering that the IMPDH of MPA-resistant Candida albicans isolates harbors Thr at the analogous position, this mutation was considered to be a marker of Pneumocystis strain selection related to MPA exposure.

The aim of this study is to strengthen these preliminary results with data from a large multicenter study.

The study will be conducted in 26 centers in France. About one hundred patients with PCP will be enrolled. Pneumocystis isolates from SOT recipients exposed to MPA and from control patients (non-SOT recipients, not exposed to MPA) will be examined.The analysis of the impdh gene was combined with a multilocus sequence typing (MLST) method (mtLSUrRNA, cytochrome b and superoxide dismutase genes) characterized by a high discriminatory power.

The expected results may show the presence of the G1020A mutation (Ala261Thr) in SOT recipients exposed to MPA and in none of the control patients not exposed to MPA. This mutation will be significantly associated with MPA exposure. It could also be associated with a specific multilocus genotype in SOT patients and none of the control patients.

The study will confirm that the G1020A mutation (Ala261Thr) represents the signature of MPA exposure. The results of the analysis of the impdh gene combined with the MLST will highlight the selection under MPA pressure of specific strains of Pneumocystis, which circulate in the population of SOT recipients.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old with PCP diagnoses, organ transplant recipient or not, acceptation to participate

Exclusion Criteria:

* < 18 years old, no acceptation to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: organ transplant recipients vs. non transplant recipient
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Presence of Pneumocystis IMPDH gene mutant or not | At patient enrollment
  The main biological parameter which will be measured will be the positive or negative result for the detection of Pneumocystis IMPDH gene mutant

CONTACTS AND LOCATIONS:
Locations (1):
- Brest University Hospital, Brest, France